CLINICAL TRIAL: NCT03866395
Title: Effects of Ivabradine on Residual Myocardial Ischemia After PCI Evaluated by Stress Echocardiography
Brief Title: Effects of Ivabradine on Residual Myocardial Ischemia After PCI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Policlinico Umberto I (Other)
Responsible Party: Principal Investigator, Massimo Mancone, (MD, PhD) Principal Investigator, Azienda Policlinico Umberto I
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04091990
Record Dates: First submitted 2018-06-01; First posted 2019-03-07 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Angina Pectoris, Stable
Keywords: Stable angina; coronary artery diseases; heart rate; exercise tolerability; diastolic function; ivabradine
MeSH Terms: conditions — Angina, Stable; Coronary Artery Disease | interventions — Ivabradine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): drug therapy according to the guidelines
- Ivabradine Group (Experimental): drug therapy according to the guidelines + Ivabradine 5 mg twice a day
  Interventions: Drug: Ivabradine

INTERVENTIONS:
Drug: Ivabradine — Ivabradine 5 mg twice a day
  Other Names: Procoralan; Corlentor
  Arms: Ivabradine Group

SUMMARY:
This is a randomized pharmacological study evaluating the effects of ivabradine in patients with residual angina after PCI. The role of ivabradine in patients with angina, without systolic dysfunction, is not yet clear. The investigators performed in all patients an echostress to evaluate the effects of therapy with ivabradine after 30 days in terms of exercise tolerance and diastolic function.

DETAILED DESCRIPTION:
BACKGROUND. Residual angina after PCI is a frequently-occurring disease. Ivabradine improves symptoms but its role in patients without left-ventricular systolic dysfunction is still unclear. The aim was to quantify the effects of ivabradine in terms of MVO2 indicators and diastolic function.

METHODS. 28 consecutive patients with residual angina after PCI were randomized to ivabradine 5 mg twice/day(IG) or standard therapy(CG). All patients performed a stress echocardiography at the enrollment and after 30 days. Myocardial oxygen consumption was estimated from: double product(DP); triple product(TP) integrating DP with ejection-time(ET). Diastolic function was evaluated determining E and A waves, E' measurements and E/E' ratio both at rest and at the peak of exercise.

ELIGIBILITY:
Inclusion Criteria:

* coronary artery disease with chronic stable angina for more than three months (Canadian Cardiovascular Society-CCS-class I-III);
* percutaneous revascularization with stent implantation at least one;
* signs/symptoms of residual ischemia; sinus rhythm; HR ≥ 70 bpm at rest;
* ability to perform an echocardiogram stress test with the tilting bicycle stress test (BST);
* good acoustic window;
* age ≥ 18 years.

Exclusion Criteria:

* drugs intolerance or hypersensitivity
* EF ≤ 40 %
* NYHA class III to IV;
* CCS IV
* atrial fibrillation or flutter
* presence of a pacemaker or implantable defibrillator
* II or III degree AV block
* HR ≤ 70 bpm at rest or sick sinus syndrome
* any condition that could interfere with the ability to exercise stress test like Wolff- Parkinson-White syndrome, left bundle branch block, left ventricular hypertrophy;
* rate-corrected QT interval (QTc) greater than 500 ms or the use of drugs that prolong the QTc interval
* symptomatic hypotension or uncontrolled hypertension (systolic blood pressure at rest ≥ 180 mmHg or diastolic blood pressure ≥ 100 mmHg)
* severe liver disease and severe renal impairment (creatinine clearance ≤ 30 ml/min)
* electrolyte disorders
* uncontrolled thyroid disease
* pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-03-05 (Actual); Primary Completion 2017-03-07 (Actual); Study Completion 2017-03-07 (Actual)

PRIMARY OUTCOMES:
Double product (DP) calculated as a product between HR and systolic blood pressure. (unit of measure: beats per minute x mmHg) | 30 days
  These, indirectly, reflect the true myocardial oxygen consumption (MVO2) and the improvement of mechanical load that the ventricle can withstand at different levels of exercise.
Triple product (TP), calculated as a product between HR, systolic blood pressure and ejection time. (unit of measure: beats per minute x mmHg x msec) | 30 days
  These, indirectly, reflect the true myocardial oxygen consumption (MVO2) and the improvement of mechanical load that the ventricle can withstand at different levels of exercise.
chronotropic reserve (unit of measure: beats per minute) | 30 days
  difference between resting heart rate and maximum heart rate at peak exercise
muscular work (unit of measure: watt) | 30 days
  These, indirectly, reflect the myocardial oxygen consumption (MVO2) and the improvement of mechanical load that the ventricle can withstand at different levels of exercise.

SECONDARY OUTCOMES:
diastolic function: PW Doppler E wave (unit of measure: cm/sec) | 30 days
  ventricular filling echocardiographic parameter
diastolic function: TDI derived E' measurements (unit of measure: cm/sec) | 30 days
  ventricular filling echocardiographic parameter. Mitral annular E' velocity was estimated as the average between lateral and septal velocity.
diastolic function: PW Doppler A wave (unit of measure: cm/sec) | 30 days
  ventricular filling echocardiographic parameter
E/E' ratio | 30 days
  ventricular filling echocardiographic parameter. TDI derived E' measurements (unit of measure: cm/sec). PW Doppler E wave (unit of measure: cm/sec)

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Mancone, Principal Investigator — Department of Cardiovascular disease, Sapienza, University of Rome, Italy
Locations (1):
- Massimo Mancone, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT03866395/Prot_SAP_000.pdf